CLINICAL TRIAL: NCT04514198
Title: Postoperative Pancreatitis and Its Correlation With Clinically Relevant Pancreatic Fistula in Pancreaticoduodenectomy- A Prospective Observational Study
Brief Title: Postoperative Pancreatitis and Its Correlation With Clinically Relevant Pancreatic Fistula in Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Dr, Asian Institute of Gastroenterology, India
Other Study IDs: POP001
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Pancreas Disease
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
AIM

To determine association between postoperative pancreatitis and pancreatic fistula

OBJECTIVES

1. To determine incidence of Clinically relevant pancreatic fistula (grade B/C) after pancreaticoduodenectomy
2. To determine role of serum amylase levels on day 1 to predict clinically relevant pancreatic fistula
3. To determine risk factors for postoperative pancreatitis and postoperative pancreatic fistula

Primaryendpoint:

Incidence of post operative pancreatitis and post operative pancreatic fistula.

Secondaryendpoints:

1. to identify the possible predictors of post operative pancreatitis.
2. to investigate the association between post operative pancreatitis and post operative pancreatic fistula.

MATERIAL AND METHODS

Study centre:

Inpatient admissions in Department of gastroenterology, Asian institute of gastroenterology, Hyderabad

Study population:

Patients who are supposed to undergo pancreaticoduodenectomy Study design: Prospective observational study

Study period:

Study will be conducted till desired sample size achieved or March 2020 to march 2022

DETAILED DESCRIPTION:
STUDY PROCEDURE:

Demographic, pathological and intraoperative data will be recorded in a prospectively maintained database populated from a combination of electronic patient records, preoperative imaging and anaesthetic charts. Preoperative clinical data included age, gender, body mass index (BMI), and the results of serum biochemical investigations including serum bilirubin, urea and amylase. The serum amylase measured throughout the study period is total amylase. Preoperative computed tomography images will beanalyzed to calculate pancreatic duct diameter at the line of transection of the pancreas anterior to the portal vein. Intraoperative data included reconstruction technique, texture of the pancreatic remnant and estimated blood loss. Blood loss data will be compiled from a combination of anaesthetic charts and perioperative blood transfusion data. Specimens will be dichotomized according to whether their pathology was associated with hard pancreatic parenchyma [pancreatic ductal adenocarcinoma (PDAC) and chronic pancreatitis] or with soft or normal pancreatic parenchyma (ampullary carcinoma, duodenal carcinoma, cholangiocarcinoma, neuroendocrine tumours and other lesions). Outcome data included length of stay in a critical care environment [defined as either an intensive care unit (ICU) or a surgical high-dependency unit (SHDU)] and length of postoperative hospital stay. All postoperative complications will be prospectively recorded and graded according to the International Study Group on Pancreatic Fistula (ISGPF) and International Study Group of Pancreatic Surgery (ISGPS) classifications and the Clavien-Dindo classification. Complications of ISGPS Grades B and C and Clavien-Dindo Grades III-V are considered clinically significant. Mortality will be recorded at 30-day and 90-day time-points.

Serum amylase will be systematically measured on POD1 and POD3 according to our institutional policy. No additional radiological or laboratory studies are required for the diagnosis of postoperative pancreatitis. No specific protocols for the treatment of POP will be followed during the study period because none are available. Due to the absence of a widely accepted definition, POP is defined according to Connor's definition1 as an elevation in serum pancreatic amylase above the upper limit of normal on postoperative day (POD) 0 or 1. At our institution, the upper limit of normal for serum pancreatic amylase is 100 U/L.

ELIGIBILITY:
Inclusion Criteria:

All patients (>18 yrs) undergoing elective Whipple's PD in Asian institute of gastroenterology, Hyderabad, Telangana.

Exclusion Criteria:

* On table inoperable patients
* Patients in cholangitis or bilirubin > 15 mg/dl
* Patients not giving consent for participation
* Patients with acute inflammatory states (cholangitis, sepsis, trauma, acute on chronic pancreatitis)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sample size : Required 35 subjects
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
To estimate incidence of Post operative Pancreatitis and post operative pancreatic fistula among patients undergoing pancreaticoduodenectomies. | 10 days
  After pancreaticoduodenectomy surgery, pancreatitis occurs it is a local inflammatory process occurring in the area of the pancreatic anastomosis after pancreas resection could induce increased systemic amylase concentration, Amylase normal range is 28--100, if it exceeds the upper normal limits it leads to post operative pancreatitis, pancreatic fistula is defined as persistent drainage of amylase rich fluid (3x > than upper limit of normal serum amylase) for greater than 3 days.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Pradeep Rebala, MBBS MS MCH, Study Chair — Asian Institute of Gastroenterology, India; Dr Shasheendra yanagandula, MBBS MS, Principal Investigator — Asian Institute of Gastroenterology, India
Locations (1):
- Asian Institute of Gastroenterology/AIG Hospitals, Hyderabad, Telangana, India

REFERENCES:
- [Derived] Shasheendra Y, Ahmed Z, Shetty MG, Hazarathaiah N, Rebala P, Rao GV. Association of Postoperative Hyperamylasemia With Clinically Relevant Postoperative Pancreatic Fistula in Pancreatoduodenectomy. Cureus. 2024 Jan 30;16(1):e53257. doi: 10.7759/cureus.53257. eCollection 2024 Jan. PMID 38435944